CLINICAL TRIAL: NCT00575068
Title: A Phase I/II Trial of Anti-CD80 Monoclonal Antibody (IDEC-114) Therapy for Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: Safety and Efficacy of IDEC-114 in the Treatment of Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114-20
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — galiximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: IDEC-114

INTERVENTIONS:
Drug: IDEC-114 — Phase 1-A Group 1 - 125 mg/m2 x 4 infusions - Study Days 1, 8, 15, 22 Phase 1-A Group 2 - 250 mg/m2 x 4 infusions - Study Days 1, 8, 15, 22 Phase 1-A Group 3 - 375 mg/m2 x 4 infusions - Study Days 1, 8, 15, 22 Phase 1-B Group 4 - 500 mg/m2 x 4 infusions - Study Days 1, 8, 15, 22 Phase II-A & II-B - Dosage start at the MTD (up to 375 mg/m2)

SUMMARY:
The purpose of this study is to determine whether anti-CD80 monoclonal antibody (IDEC-114) is effective in the treatment of follicular B-cell non-Hodgkin's lymphoma. This drug has never been studied in patients with lymphoma, however, it has been studied in psoriasis patients at various dose levels and schedules.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma that has relapsed or has failed primary therapy
* Progressive disease requiring further treatment
* Bidimensionally measurable disease
* Acceptable hematologic status
* Prestudy WHO performance status of 0, 1, or 2
* Expected survival of >/= 3 months
* Patients with reproductive potential must follow accepted birth control methods during treatment and for 3 months after completion of treatment
* Female patients must not be pregnant or lactating
* Recovered fully from any significant toxicity associated with prior surgery, radiation treatments, chemotherapy, biological therapy, ABMT, or investigational drugs

Exclusion Criteria:

* Cancer radiotherapy, biological therapy, or chemotherapy within 3 weeks of first scheduled treatment (6 weeks if nitrosourea or mitomycin-C)
* Prednisone or other immunosuppressive therapy within 3 weeks of first scheduled treatment
* Prior antibody therapy for lymphoma (including radioimmunotherapy) within 6 months prior to first scheduled treatment
* Previous exposure to IDEC-114 or any anti-CD80 antibody
* ABMT within 6 months prior to first scheduled treatment
* Abnormal liver function
* Abnormal renal function
* Presence of chronic lymphocytic leukemia (CLL)
* Presence of CNS lymphoma
* Presence of HIV infection or AIDS
* Prior diagnosis of aggressive non-Hodgkin's lymphoma or mantle-cell lymphoma
* Another primary malignancy (other than squamous cell and basal cell carcinoma of the skin, in situ carcinoma of the cervix, or treated prostate cancer with a stable PSA) for which the patient has not been disease-free for at least 3 years
* Serious nonmalignant disease which would compromise protocol objectives in the opinion of the investigator and/or the sponsor
* New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to first scheduled treatment
* Major surgery, other than diagnostic surgery, within 4 weeks prior to first scheduled treatment
* Pleural invasion and/or effusion with positive cytology for lymphoma
* Peritoneal invasion and/or ascites with positive cytology for lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2002-01; Primary Completion 2002-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To characterize the safety profile of IDEC-114 and to define their duration and reversibility | March 2010

SECONDARY OUTCOMES:
To evaluate PK | March 2010
To monitor presence of human anti galiximab antibody | March 2010
To evaluate efficacy | March 2010
To identify Nk functional assays that may predict galiximab efficacy | March 2010

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Tucson, Arizona
  - Research Site, Rochester, Minnesota
  - Research Site, Buffalo, New York
  - Research Site, Durham, North Carolina